CLINICAL TRIAL: NCT06430918
Title: Coexistence of Night Pain and Neuropathic Pain in Patients With Knee Osteoarthritis
Brief Title: Neuropathic Pain and it's Relation to Sleep Quality in Knee Osteoarthritis
Status: Enrolling by invitation | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Taciser Kaya, MD, Professor, Bozyaka Training and Research Hospital
Other Study IDs: 226092BK
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Sleep Disturbance; Neuropathic Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Parasomnias; Neuralgia | interventions — Restraint, Physical; Surveys and Questionnaires; Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis: Knee OA patients diagnosed according to the ACR Classification Criteria
  Interventions: Other: physical examination, questionnaires and inventories

INTERVENTIONS:
Other: physical examination, questionnaires and inventories — Questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed.
  Other Names: Questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed.

SUMMARY:
The primary aim is to investigate the frequency and severity of neuropathic pain and its association with night pain in patients with knee osteoarthritis. For this purpose a progressive longitudinal study design was planned. The secondary aim is to investigate the relationship between night pain and neuropathic pain and sleep quality.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis in the world. Classically, OA presents with joint pain and loss of function; however, the disease is clinically very variable and can present merely as an asymptomatic incidental finding to a devastating and permanently disabling disorder.

The severity of knee pain caused by osteoarthritis, often does not correlate with the degree of degenerative changes in the joint. In patients reporting night pain, this may be related to inflammation, but in the absence of clinical and laboratory findings of inflammation, it is not possible to explain night pain only by the degree of joint damage. The existence of a relationship between night pain and neuropathic pain may be a guide in looking for neuropathic pain in patients who have night pain and experience this pain severely and thus for planning an appropriate treatment for the patient.

Patients with stage 2-4 knee OA will be evaluated in terms of demographic variables and outcome measurement parameters specified in the case report form. The relationship between neuropathic pain scores and knee pain severity will be sought. It will be studied whether there is a difference in outcome measurement parameters between those with neuropathic pain and those without. Correlation analysis will be performed between sleep quality score and pain intensity scores. The determinants of sleep quality will be evaluated by regression analysis.

American College of Rheumatology criteria will be recruited. Demographics and disease related variables will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Having a clinical diagnosis of knee osteoarthritis according to the American Rheumatology Association/ACR criteria 2. Knee OA is of Kellgren-Lawrence stage 2-4 3. The participant gives signed consent

-

Exclusion Criteria:

Exclusion Criteria:

1. Having diabetes mellitus 2. Chronic kidney failure 3. Hypothyroidism 4. Presence of orthopedic disability (such as implant, prosthesis, contracture, shortness) in the lower extremity 4. Neurological diseases that can cause neuropathic pain 5. Presence of fibromyalgia 6. Malignancy 7. Pregnancy 8. Neurological deficit in the lower extremity 9. Drug use that may cause neuropathy (colchicine, etc.) İn the last 3 months 10. Drug use (antidepressant, antipsychotic, antiepileptic) due to sleep disturbance or widespread pain in the last 3 months.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 2-4 knee OA will be evaluated in terms of demographic variables and outcome measurement parameters specified in the case report form.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain; 4 Questions Neuropathic Pain Questionnaire | through study completion, an average of 1 year
  The DN4 questionnaire (4 Questions Neuropathic Pain Questionnaire) will be used. It is a clinician-administered questionnaire. It consists of ten items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient. Three items are based on the clinical examination. The clinician assesses whether there is reduced sensation (hyposthesia) to touch or pinprick and whether light brushing increases or causes pain (allodynia). All of the positive items are scored as one point and total score is sum of the scores of these positive items. The diagnosis is based on 4/10 cut-off value.

SECONDARY OUTCOMES:
Sleep quality | through study completion, an average of 1 year
  Jenkins Sleep Scale.The four-item questionnaire evaluates the frequency and intensity of certain sleep difficulties in respondents. Questions queries the number of days in which the patient was subjected to sleep problems. The maximum possible score is 20 and higher scores indicate much more sleep disturbance. A mean score of two or more is considered as sleep disturbance presence.
Depression and Anxiety; The Hospital Anxiety and Depression Scale (HADS) | through study completion, an average of 1 year
  The Hospital Anxiety and Depression Scale (HADS) was developed by Zigmond and Snaith in 1983. It is used to detect whether the patient is in the depressive or anxious status. It is not a diagnostic tool but gives to physician an idea about the patient's emotional status. It consists of fourteen items. Seven items are related to anxiety and the other seven depression
Quality of life level; KOOS (KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) "Quality of Life" subgroup | through study completion, an average of 1 year
  KOOS evaluates the symptoms and functional problems related to knee OA and knee injury. It consists of five subscales. In this study authors intended to assess the life quality by using the quality of life level subscale of this scale.
Disability; KOOS (KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) "Activities of Daily Life and Function" subgroup | through study completion, an average of 1 year
  Disability; KOOS (KNEE INJURY AND OSTEOARTHRITIS OUTCOME SCORE) "Activities of Daily Life and Function" subgroup
Night pain (VAS, 0-10 cm) Participants will be asked to report the pain intensity that they feel on a line between 0 and 10, higher scores indicating more intense pain. | through study completion, an average of 1 year
  Participants will be asked to report the pain intensity that they feel on a line between 0 and 10, higher scores indicating more intense pain.

CONTACTS AND LOCATIONS:
Overall Officials: Taciser Kaya, Prof., Principal Investigator — Izmir Bozyaka Training and Research Hospital İzmir, Turkey; Berna Kirilmaz Colak, MD, Principal Investigator — Izmir Bozyaka Training and Research Hospital İzmir, Turkey; Bugra Ince, Assoc. prof., Principal Investigator — Izmir Bozyaka Training and Research Hospital İzmir, Turkey
Locations (1):
- Izmir Bozyaka Training and Reseach Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Hoper J, Schraml L, Gierthmuhlen J, Helfert SM, Rehm S, Hartig S, Schroder O, Lankes M, Traulsen FC, Seekamp A, Baron R. Changes of Somatosensory Phenotype in the Course of Disease in Osteoarthritis Patients. Int J Environ Res Public Health. 2020 Apr 29;17(9):3085. doi: 10.3390/ijerph17093085. PMID 32365479
- [Result] Wylde V, Palmer S, Learmonth ID, Dieppe P. Somatosensory abnormalities in knee OA. Rheumatology (Oxford). 2012 Mar;51(3):535-43. doi: 10.1093/rheumatology/ker343. Epub 2011 Nov 24. PMID 22120461